CLINICAL TRIAL: NCT05007496
Title: Phase II Randomized Double Blind Clinical Trial Three Preventive Vaccine Formulations Consisting of Autologous Dendritic Cells and Lymphocytes Incubated With Different Quantities of Spike Protein Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2), in Subjects Not Proven Actively Infected or Never Infected With COVID-19
Brief Title: Preventive Dendritic Cell Vaccine, AV-COVID-19, in Subjects Not Actively Infected With COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Aivita Biomedical, Inc. (Industry)
Collaborators: PT AIVITA Biomedika Indonesia (Unknown); Kariadi Hospital (Unknown); Central Army Hospital RSPAD Gatot Soebroto (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: CL-COV-P02-ID
Record Dates: First submitted 2021-08-11; First posted 2021-08-16 (Actual); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: COVID-19
Keywords: Prevention
MeSH Terms: conditions — COVID-19 | interventions — AV-COVID-19 vaccine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AV-COVID-19 (0.1 mcg S-protein) (Experimental): DCL previously incubated with 0.1 mcg spike protein
  Interventions: Biological: AV-COVID-19
- AV-COVID-19 (0.33 mcg S-protein) (Experimental): DCL previously incubated with 0.33 mcg spike protein
  Interventions: Biological: AV-COVID-19
- AV-COVID-19 (1.0 mcg S-protein) (Experimental): DCL previously incubated with 1.0 mcg spike protein
  Interventions: Biological: AV-COVID-19

INTERVENTIONS:
Biological: AV-COVID-19 — DCL previously loaded with varying quantity of S-protein

SUMMARY:
This is a phase 2 randomized, double-blind clinical trial testing an anti-SARS-CoV-2 COVID-19 vaccine (AV-COVID-19) made on site using PT AIVITA Biomedika Indonesia's vaccine-enabling kit for the prevention of COVID-19 infection. The product is a subject-specific personal vaccine that consists of autologous dendritic cells and lymphocytes (DCL) previously incubated with a quantity of SARS-CoV-2 spike protein (S-protein) which was shown to be safe in a phase 1 study also conducted in Indonesia. In this phase 2 study, efficacy is assessed via enhanced S-protein-specific T-cell response by comparing results before and after vaccination. Safety is confirmed via laboratory values, observation and regular patient reporting.

DETAILED DESCRIPTION:
In this phase 2 study, a single dose of AV-COVID-19 DCL vaccine is injected subcutaneously in the forearm (left or right) at week 0 (day-0), to facilitate inspection and avoid confusion of local post-injection reactions or shoulder pain. Follow-up visits to assess safety are performed at 1, 2, and 4 weeks after vaccination, with laboratory safety tests performed at weeks 1 and 4, and only at week 2 if any clinically significant changes at screening up to week 1. At each visit, the injection site is assessed, and the subject is asked about symptoms, and at weeks 0 (baseline before injection), 2 and 4, blood is drawn for immunogenicity testing. Reaction data at the injection site and safety profile are obtained by telephone to subjects on days 1, 2, and 3 after vaccine injection. Subjects are asked specifically about local injection site reactions and systemic flu-like symptoms (fever, chills, muscle aches, joint pain) for 7 days after injection. Adverse events (AE) are collected for 28 days after injection. Evaluation of laboratory tests for clinical safety parameters are carried out at screening as well as immediately before vaccination and on day 7 and day 28 post-vaccination. Serious adverse events (SAE), recent medical conditions, and other events requiring medical intervention are recorded for 2 months after vaccination. Vaccine enabling kits are made by PT AIVITA Biomedika Indonesia. All vaccines are made in Indonesia on site at participating hospitals and clinical sites.

ELIGIBILITY:
Inclusion Criteria:

* Understands and agrees to comply with research procedures and provides written informed consent
* Physical and mental health meet criteria to participate, which includes factors associated with increased risk of exposure to SARS-CoV-2, such as age > 65, mild to moderate obesity (BMI 30-40), hypertension controlled with medication, drug controlled hyperlipidemia, diabetes controlled with medication, mild chronic lung disease
* Vein access permits for blood collection
* For people with reproductive ability, adequate contraception and negative pregnancy test for women

Exclusion Criteria:

* Have active symptoms of COVID-19 infection
* Diagnosed with COVID-19 with a positive PCR test in the past 3 months
* Positive SARS-CoV-2 rapid antibody IgG test
* Positive pregnancy test
* Known to have immunodeficiency disease
* Are taking immunosuppresive drugs and/or corticosteroids in the long term
* Have a condition requiring oxygen supplementation
* Previously diagnosed with invasive cancer and receiving anti-cancer therapy in addition to hormonal therapy for breast or prostate cancer
* History of thromboembolism or genetic predisposition to thromboembolism, or being on anti-thromboembolic therapy other than low-dose aspirin
* Physical or mental disability that prevents you from carrying out normal daily activities
* In the Investigator's judgement, have illnesses or medical conditions that could preclude participation
* Excessive obesity: BMI > 40
* Uncontrolled hypertension: systolic > 180, diastolic > 100
* Not willing to sign written consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2021-04-14 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Efficacy based on T-cell-induced immune response | 4 weeks
  ELISPOT assay at baseline, week 2 and week 4 post-vaccination

SECONDARY OUTCOMES:
Adverse event frequency and incidence | 4 weeks
  Confirm safety of AV-COVID-19 via laboratory values and adverse event reporting from baseline to 28-days post-vaccination
Optimal formulation | 4 weeks
  Choose the optimal formulation (0.1, 0.33, 1.0 mcg S-protein)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Jonny, SpPD-KGH, MKes, MM, Principal Investigator — Rumah Sakit Pusat Angkatan Darat Gatot Soebroto
Locations (1):
- RSPAD Gatot Soebroto, Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided